CLINICAL TRIAL: NCT06826898
Title: A Prospective, Single-center, Randomized, Evaluator/subject-blinded, Controlled Clinical Study: to Evaluate the Effectiveness of the Use of a Novel Crosslinking Hyaluronan Hydrogel on the Prevention of the Adhesion Occurrence After Anterior Talofibular Ligament Repair Surgery
Brief Title: To Evaluate the Effectiveness of the Use of a Novel Crosslinking Hyaluronan Hydrogel on the Prevention of the Adhesion Occurrence After Anterior Talofibular Ligament Repair Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Talent Cro Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDCT-SCDH
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Anterior Talofibular Ligament Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Absorbable Adhesion Barrier (Experimental): DEFEHERE Absorbable Adhesion Barrier, 1.0 mL/syringe
  Interventions: Device: DEFEHERE Absorbable Adhesion Barrier
- Sham (Sham Comparator): conventional therapy without using any antiadhesion product
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: DEFEHERE Absorbable Adhesion Barrier — DEFEHERE Absorbable Adhesion Barrier, 1.0 mL/syringe
  Arms: Absorbable Adhesion Barrier
Device: Sham (No Treatment) — conventional therapy without using any antiadhesion product
  Arms: Sham

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of the use of a novel crosslinking hyaluronan hydrogel on the prevention of the adhesion occurrence after anterior talofibular ligament repair surgery. With applying crosslinking hyaluronan hydrogel, the range of motion (ROM) of the ankle is expected to be better than sham group.

ELIGIBILITY:
Inclusion Criteria:

1.1 Voluntarily participate and sign an informed consent form; 1.2 Age 18 to 60 years of male or female; 1.3 Patients experiencing lateral ankle pain discomfort, confirmed by MRI to have anterior talofibular ligament (ATFL) injury; 1.4 History of recurrent ankle inversion sprains three times or more, with no improvement after six months of conservative treatment, and scheduled for ATFL repair surgery; 1.5 Willing to comply with all follow-up requirements of the trial protocol.

Exclusion Criteria:

2.1 Severe ankle osteoarthritis; 2.2 Patients with a history of ankle fracture or surgery; 2.3 Undergoing foot- or ankle-related treatments that may affect the trial results; 2.4 Presence of skin infection, skin defects, or need for skin grafting at the surgical site; 2.5 Uncontrolled chronic diseases, such as diabetes mellitus; 2.6 Presence of autoimmune diseases (such as Autoimmune Collagenopathy, rheumatoid arthritis), malignancies, coagulation disorders, heart diseases, psychiatric illnesses, or other conditions that may pose higher risks to patients in the trial; 2.7 Use of corticosteroids within the past 6 months, systemic corticosteroids within the past month, immunosuppressive drugs within the past 3 months, or daily use of non-steroidal anti-inflammatory drugs (NSAIDs) within the past week, or occasional use within 8 hours (patients using nasal/inhaled corticosteroids may be considered for inclusion) ; 2.8 Clinically significant coagulation abnormalities or undergoing anticoagulant therapy within 10 days before surgery or currently taking anticoagulant drugs; 2.9 Known allergy to sodium hyaluronate or any components of medical devices;allergy to Gram-positive bacterial protein or streptococcal protein；or other severe allergic history deemed unsuitable for participation by the investigators; 2.10 Pregnant, lactating women, or women planning to become pregnant during the trial period; 2.11 Other conditions deemed unsuitable for participation by the investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Range of Motion (ROM) | day 14
  Measure the range of plantar flexion, dorsiflexion, inversion, and eversion of the ankle.

SECONDARY OUTCOMES:
Range of Motion (ROM) | baseline, day 28, 49, 70
  Measure the range of plantar flexion, dorsiflexion, inversion, and eversion of the ankle.
Anterior Talar Translation (ATT) | baseline, day 14, 28, 49, 70
  On the sagittal plane, the talus below the tibia will be pulled forward to test the integrity of the anterior talofibular ligament.
Visual Analogue Scale (VAS) for pain | baseline, day 14, 28, 49, 70
  The VAS scale uses a 10 cm line labelled at '0' with 'no pain' and '10' with 'worst pain'
Cumberland Ankle Instability Tool (CAIT) questionnaire | baseline, day 14, 28, 49, 70
  The Cumberland Ankle Instability Tool (CAIT) is a 9-item 30-point scale that measures the severity of functional ankle instability.
American Orthopedic Foot and Ankle Society (AOFAS) questionnaire | baseline, day 14, 28, 49, 70
  AOFAS includes 9 items that can be divided into three subscales (pain, function and alignment).
Foot and Ankle Ability Measure (FAAM) questionnaire | baseline, day 14, 28, 49, 70
  A self-report outcome instrument developed to assess physical function for individuals with foot and ankle related impairments. The FAAM is a 31-item questionnaire divided into two subscales: Activities of Daily Living Subscale and Sports Subscale.
Subject self-assessment satisfaction scores | day 14, 28, 49, 70
  Subject self-assessment satisfaction scores

CONTACTS AND LOCATIONS:
Locations (1):
- Show Chwan Memorial Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided